CLINICAL TRIAL: NCT00660322
Title: Using the Telephone to Improve Care in Childhood Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Jane Garbutt, MB,ChB, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HS015378
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Asthma
Keywords: Asthma; Telemedicine; Randomized controlled trial
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Families assigned to the control arm will receive usual asthma care from the child's primary care provider.
- Intervention (Experimental): The Telephone Asthma Program and usual care.
  Interventions: Behavioral: Telephone Asthma Program

INTERVENTIONS:
Behavioral: Telephone Asthma Program — The parent will have access to a trained asthma coach for 12 months. The coach will call the parents at mutually convenient times (up to 12 times a year) to work on 4 targeted asthma behaviors:
  1. Using asthma controller medications as prescribed
  2. Having and Asthma Action Plan available to all who may need it.
  3. Using asthma rescue medications with the child's first symptoms.
  4. Having a collaborative relationship with the child's primary care provider that includes asthma check-ups at least twice a year.
  Arms: Intervention

SUMMARY:
Asthma is the most common chronic disease of childhood and a major cause of morbidity in the United States. If asthma symptoms are controlled, a child with asthma can stay well and lead a normal life. Daily use of inhaled steroids controls symptoms and reduces morbidity and emergent health care utilization in children with persistent asthma, and is safe for long-term use. However, inhaled steroids are underused in community asthma care.

The Telephone Asthma Program (TAP) is a series of brief, telephone calls with a trained coach to help the parent manage the child's asthma care. The coach will teach self-management skills, help the parent to use the child's asthma medicines effectively, provide support and remind the parent to go for follow-up care with the pediatrician. We hypothesized that the Telephone Asthma Program will reduce the incidence of acute exacerbations of asthma that require emergent care, improve the quality of life of children with asthma and their parents, and increase the daily use of inhaled steroids in children with persistent asthma. We evaluated the Telephone Asthma Program in a randomized controlled trial involving 362 children aged 5 to 12 years old cared for by community pediatricians. Eligible children were randomized to the TAP program or usual care by their pediatrician.

DETAILED DESCRIPTION:
Asthma morbidity is largely preventable with effective maintenance care. National guidelines recommend 1) daily treatment with inhaled corticosteroids (ICS) to prevent asthma symptoms and activity limitations, minimize acute exacerbations and maintain normal lung function; 2) early intervention guided by a written Asthma Action Plan for worsening symptoms;3) a partnership between the primary care provider, the patient and their family to develop shared treatment goals, select an appropriate treatment plan, resolve asthma-related concerns, and provide support for day-to-day care, and 4) periodic assessments (every 1 to 6 months) by the physician to monitor asthma control and assess if the goals of therapy are being met, with asthma self-management education provided at diagnosis and reinforced at every opportunity. Despite widespread dissemination of these guidelines, under-use of controller medications is pervasive, home management of an acute exacerbation is often delayed and inadequate, and only 50% of asthmatic children report maintenance care visits twice a year. Most primary care pediatricians do not provide education about use of preventive treatments or self-management behaviors citing lack of confidence in their ability to effect change, logistical issues such as lack of time, educational materials, support staff, and inadequate reimbursement as significant barriers to these activities. Practical, efficient interventions to improve maintenance asthma care in office-practice are needed.

In response to complaints from community pediatricians in our practice-based research network that few children with persistent asthma used their controller medications as prescribed we collaborated with local asthma experts and the telephone triage service at our children's hospital to develop and evaluate a 12-month telephone-coaching program to provide education and support to parents to improve asthma self-management for their children. The Telephone Asthma Program (TAP) was provided in addition to usual care, and was evaluated in a randomized controlled trial (RCT).

The TAP program was based on the Transtheoretical Model of Behavior Change developed by James Prochaska. This model postulates a series of 5 ordered stages of readiness to change to a desired behavior (Precontemplation, Contemplation, Preparation, Action and Maintenance). The desired behaviors for TAP were: 1) using controller medications as prescribed, 2) administering rescue medications at the child's first signs of an asthma exacerbation, 3) having an up-to-date asthma action plan readily available for all who may need it, and 4) having a collaborative relationship with the child's PCP that included regular asthma check-up visits at least every 6 months. Our goal was that all 4 behaviors would be addressed by the coach for each parent throughout the 12-month program period. Guided by computerized telephone protocols the coach provided tailored care advice appropriate for the parent's stage of readiness for behavior change. In this way, the coach could provide education and support to help the parent to provide effective asthma care at home for their child, and supplement the care provided by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma for at least a year
* At least one acute exacerbation of asthma in past 12 months that required a visit to the emergency department, hospitalization or an unscheduled office visit for acute care and/or a course of oral steroids.
* Taking daily controller medications or symptoms consistent with persistent asthma

Exclusion Criteria:

* No phone
* Unable to speak English
* Child has another disease that requires regular monitoring by pediatrician
* A sibling is already enrolled in the study
* Child's primary asthma provider is an asthma specialist

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 362 (Actual)
Dates: Start 2004-01; Primary Completion 2006-01 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Parental asthma-related quality of life | one year
Urgent care events for asthma | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jane Garbutt, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Garbutt J, Bloomberg G, Banister C, Sterkel R, Epstein J, Bruns J, Swerczek L, Wells S. What constitutes maintenance asthma care? The pediatrician's perspective. Ambul Pediatr. 2007 Jul-Aug;7(4):308-12. doi: 10.1016/j.ambp.2007.03.007. PMID 17660103
- [Derived] Garbutt JM, Banister C, Highstein G, Sterkel R, Epstein J, Bruns J, Swerczek L, Wells S, Waterman B, Strunk RC, Bloomberg GR. Telephone coaching for parents of children with asthma: impact and lessons learned. Arch Pediatr Adolesc Med. 2010 Jul;164(7):625-30. doi: 10.1001/archpediatrics.2010.91. PMID 20603462